CLINICAL TRIAL: NCT05161572
Title: A Randomized Phase II Trial of Perioperative Chemoimmunotherapy Verses Perioperative Chemoimmunotherapy Plus Preoperative Chemoradiation for Locally Advanced Gastric (G) or Gastroesophageal Junction (GEJ) Adenocarcinoma
Brief Title: Perioperative Chemoimmunotherapy With/Without Preoperative Chemoradiation for Locally Advanced Gastric Cancer
Acronym: NeoRacing
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficult in recruiting participants
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhen Zhang, Director of the department of radiation oncology, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDRT- LAGCCS004
Record Dates: First submitted 2021-11-21; First posted 2021-12-17 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Stomach Neoplasms; Esophagogastric Junction Disorder; Neoadjuvant Therapy; Chemoradiotherapy; Immunotherapy; Gastrectomy; Adenocarcinoma; Adjuvant Therapy
Keywords: Locally advanced gastric cancer; Gastroesophageal junction adenocarcinoma; Perioperative chemotherapy; Preoperative chemoradiation; PD-1 antibody
MeSH Terms: conditions — Stomach Neoplasms; Adenocarcinoma | interventions — Oxaliplatin; tegafur-gimeracil-oteracil; sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Perioperative chemotherapy plus PD-1 antibody plus preoperative chemoradiotherapy (Experimental): In this arm, patients will receive preoperative chemoradiotherapy (45Gy/25Fractions), two cycles of SOX and three cycles of PD-1 antibody, followed by D2 surgery and three more cycles of SOX and PD-1 antibody. Then PD-1 antibody will be given until one year after surgery.
  Interventions: Drug: Oxaliplatin; Drug: Tegafur-Gimeracil-Oteracil; Drug: Sintilimab; Radiation: Concurrent chemoradiation; Procedure: D2/R0 gastrectomy
- Perioperative chemotherapy plus PD-1 antibody (Experimental): In this arm, patients will receive three cycles of SOX and PD-1 antibody, followed by D2 surgery and three more cycles of SOX and PD-1 antibody. Then PD-1 antibody will be given until one year after surgery.
  Interventions: Drug: Oxaliplatin; Drug: Tegafur-Gimeracil-Oteracil; Drug: Sintilimab; Procedure: D2/R0 gastrectomy

INTERVENTIONS:
Drug: Oxaliplatin — The SOX regimen consists of S-1 and oxaliplatin and is repeated every three weeks. Oxaliplatin will be administered intravenously at 130 mg/m2 on day 1.
Drug: Tegafur-Gimeracil-Oteracil — The SOX regimen consists of S-1 and oxaliplatin and is repeated every three weeks. S-1 is administered orally at 40-60 mg twice a day for 14 consecutive days. Then, the patients will have a one-week rest period. The dose of S-1 is according to the body-surface area (BSA): patients with a BSA of less than 1.25 m2 receive 80 mg daily; those with a BSA of 1.25 m2 or more but less than 1.5 m2 receive 100 mg daily; and those with a BSA of 1.5 m2 or more receive 120 mg daily.
Drug: Sintilimab — The immunotherapy includes perioperative treatment and postoperative maintenance treatment. The PD-1 mAb used will be sintilimab, and the dose is 200 mg intravenously every three weeks. Regardless of which arm, the courses of immunotherapy that will be received by the enrolled patients are the same: 3 times preoperatively, 3 times postoperatively, and then maintained until one year after surgery.
Radiation: Concurrent chemoradiation — The radiotherapy (RT) consists of 45 Gy delivered in 25 fractions every five days per week for five weeks. The dose of concurrent ChT is 60 mg/m2 S-1 orally, oral tablets twice daily, days 1-5 of each week.
  Arms: Perioperative chemotherapy plus PD-1 antibody plus preoperative chemoradiotherapy
Procedure: D2/R0 gastrectomy — Gastrectomy with standard D2 lymphadenectomy is recommended. The type of gastrectomy performed depends on the location and extent of the primary lesion. For GEJ or upper third tumors, a 3 cm esophageal margin is recommended, and a total gastrectomy or esophagogastrectomy is performed. For middle third tumors, the gastric margin is recommended to be more than 5 cm, and a total gastrectomy is performed. For lower third tumors, a 2 cm duodenal margin is recommended, and a subtotal or total gastrectomy is performed. Billroth I or Roux-en-Y gastrojejunostomy is performed for distal gastrectomy patients. Roux-en-Y esophagojejunostomy is performed for patients receiving total gastrectomy.

SUMMARY:
NeoRacing is a randomized phase II trial carried out at Fudan University Shanghai Cancer Center (FUSCC) in China. The study can be divided into the screening stage, treatment stage and follow-up stage. The enrolled patients will receive perioperative SOX chemotherapy, PD-1 antibody (sintilimab) and radical surgery, with or without preoperative CRT. The patients were randomized by stratified permutated block randomization on a web-based system . The status of peritoneal cytological examination (CY0 vs. CY1) was the stratification factor. The study protocol was approved by the Ethics Committee of FUSCC. All patients provided written informed consent before recruitment. Monitoring will be carried out in this tri

DETAILED DESCRIPTION:
Perioperative chemotherapy (ChT) and preoperative chemoradiation (CRT) are both the standard treatments for locally advanced gastric cancer (LAGC). CRT can achieve a higher pathological complete regression (pCR) rate, but whether this higher pCR rate can be transformed into a long-term survival benefit remains inconclusive. Therefore, relevant studies are in progress. On the other hand, immunotherapy has been established for the first-line treatment of advanced gastric cancer (AGC) and has been widely explored in the perioperative setting. The combination of chemotherapy/radiotherapy and immunotherapy may have a synergistic effect, which will lead to a better antitumor effect. The preliminary reports of ongoing studies show promising results, including a further improved pCR rate. However, the preferred treatment combination for LAGC is still not established. To solve this problem, we are carrying out this randomized phase II trial, which aims to evaluate the efficacy and safety of perioperative chemotherapy plus the use of PD-1 antibodies with or without preoperative chemoradiation for LAGC.

Perioperative chemotherapy (ChT) and preoperative chemoradiation (CRT) are both the standard treatments for locally advanced gastric cancer (LAGC). CRT can achieve a higher pathological complete regression (pCR) rate, but whether this higher pCR rate can be transformed into a long-term survival benefit remains inconclusive. Therefore, relevant studies are in progress. On the other hand, immunotherapy has been established for the first-line treatment of advanced gastric cancer (AGC) and has been widely explored in the perioperative setting. The combination of chemotherapy/radiotherapy and immunotherapy may have a synergistic effect, which will lead to a better antitumor effect. The preliminary reports of ongoing studies show promising results, including a further improved pCR rate. However, the preferred treatment combination for LAGC is still not established. To solve this problem, we are carrying out this randomized phase II trial, which aims to evaluate the efficacy and safety of perioperative chemotherapy plus the use of PD-1 antibodies with or without preoperative chemoradiation for LAGC.

The results of the NeoRacing study will provide important information concerning the application of PD-1 antibodies in LAGC patients during the preoperative setting. Meanwhile, the two treatment protocols will be compared in terms of efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically confirmed gastric adenocarcinoma (G) or gastroesophageal junction adenocarcinoma (GEJ, excluding Siewert type I).
2. The clinical stage of the enrolled patients was cT3-4aN+M0 or cT4bNanyM0. Patients with a CY1 status but no other distant metastasis were allowed for patient recruitment. The clinical stage of CY1 patients is cT3-4aN+M1 (CY1 only) or cT4bNanyM1 (CY1 only) (the 8th AJCC staging system of GC).
3. The tumor was considered to be potentially resectable, which was verified by a multidisciplinary team including a surgical investigator.
4. At least one evaluable lesion on abdominal CT/MRI according to the RESIST 1.1 protocol is required.
5. An ECOG (Eastern Cooperative Oncology Group) performance status of 0-1.
6. The patient's physical state and organ function can tolerate the planned treatment of the study protocol, including perioperative chemotherapy with the SOX regimen and immunotherapy with PD-1 monoclonal antibody, preoperative concurrent chemoradiotherapy (45 Gy/25 fractions/S-1), and major abdominal surgery.
7. The baseline laboratory examinations of the patients met the following criteria:

   1. An adequate hematological function: an absolute neutrophil count (ANC) ≥ 1.5×109/L; a platelet count ≥ 100×109/L; a hemoglobin level ≥ 90 g/L.
   2. Adequate liver function: total bilirubin ≤ 1.5×upper limit of normal (ULN); AST/ALT < 2.5×ULN; ALP ≤ 2.5×ULN; ALB ≥ 30 g/L.
   3. Adequate renal function: serum creatinine ≤ 1.5 × ULN; creatinine clearance rate ≥ 60 ml/min.
   4. Adequate coagulation function: INR/PT ≤ 1.5×ULN; APTT ≤ 1.5×ULN.
8. There was no serious concomitant disease, and the patient's life expectancy was more than 6 months.
9. Male or female. Age ≥ 18 years and ≤ 75 years.
10. Patients agreed to sign a written informed consent before recruitment.
11. Patients had good compliance with the study procedures, including laboratory examinations, auxiliary examinations and treatment.
12. The female patients should not be pregnant or breastfeeding.
13. The female patients agreed to take contraceptive measures during the treatment and within 120 days after the last dose of PD-1 mAb or 180 days after the last dose of chemotherapy or radiotherapy.

Exclusion Criteria:

1. Clinical or histopathological evidence of peritoneal seeding (P1) or distant metastasis (M1).
2. Patients who have previously received surgery, chemotherapy, radiotherapy or immunotherapy for gastric cancer.
3. Patients had a history of cancer in the five years before randomization except for squamous or basal cell carcinoma of the skin that had been effectively treated and superficial bladder cancer, cervical carcinoma in situ and breast cancer in situ that had been treated by surgery.
4. Pregnant or lactating females or planning to become pregnant or lactating.
5. History of allergy to any drugs involved in this study.
6. History of allogeneic stem cell transplantation or organ transplantation.
7. Vaccinated with a live vaccine within 4 weeks before recruitment.
8. History of anti-PD-1, PD-L1, PD-L2 or any other specific T cell costimulation or checkpoint pathway targeted therapy.
9. History of using steroids (dose > 10 mg/d prednisone) or other systemic immunosuppressive therapy within 14 days before recruitment, except for patients treated with the following regimen: steroids used for hormone replacement (dose > 10 mg/d prednisone); local application of steroids with little systemic absorption; short-term (≤ 7 days) use of steroids to prevent allergy or vomiting.
10. Patients with weight loss of more than 20% within 2 months before recruitment.
11. Uncontrolled systemic diseases, including diabetes and hypertension.
12. Failure of important organs (heart, lung, liver, kidney, etc.).
13. Moderate or severe renal injury [creatinine clearance ≤ 50 ml/min (according to Cockroft & Gault equation)] or SCR > ULN.
14. Dipyrimidine dehydrogenase (DPD) deficiency.
15. Patients with central nervous system (CNS) disorders, peripheral nervous system disorders or psychiatric diseases.
16. A cerebrovascular accident that occurred within 6 months before recruitment.
17. Patients with a known history of uncontrolled or symptomatic angina, uncontrolled arrhythmias and hypertension, congestive heart failure, cardiac infarction within 6 months prior to study recruitment, or cardiac insufficiency.
18. Patients who have the following history of pulmonary diseases: interstitial lung disease, noninfectious pneumonia, pulmonary fibrosis, acute lung disease, or pulmonary embolism.
19. Patients with severe gastrointestinal bleeding, gastrointestinal perforation, or gastrointestinal fistula and patients who cannot swallow to take the drug orally.
20. Patients with upper gastrointestinal obstruction, dysfunction or malabsorption syndrome that can affect the absorption of oral chemotherapy drugs.
21. Uncontrollable pleural effusion, pericardial effusion, or ascites that occurred within two weeks before recruitment.
22. Patients with a history of active autoimmune disease or refractory autoimmune disease.
23. Severe chronic or active infections requiring systemic antibiotics, antifungal or antiviral therapy, including tuberculosis and AIDS.
24. Known history of human immunodeficiency virus (HIV) infection.
25. Patients with untreated chronic hepatitis B or HBV-DNA exceeding 500 IU/ml or HCV-RNA positivity.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Pathological complete regression (pCR) rate | 6 months after the enrollment of the last subject
  The primary endpoint is the pathological complete regression (pCR) rate: the proportion of patients who achieve pCR after preoperative therapy. Patients with a CY0 status at the time of enrollment should have no residual tumor cells in the primary lesion and in the dissected lymph nodes in the surgical specimens (ypT0N0M0). Patients with a CY1 status at the time of enrollment should reach both ypT0N0M0 and a CY0 status.

SECONDARY OUTCOMES:
Pathological response rate (pRR) | 6 months after the enrollment of the last subject
  1) The pathological response rate (pRR) is defined as the proportion of patients with a pathological response. The tumor regression will be evaluated according to Ryan's tumor regression grading (TRG). The pathological response is defined as TRG0 and TRG1 of the primary lesion after preoperative therapy.
R0 resection rate | 6 months after the enrollment of the last subject
  The R0 resection rate is defined as the proportion of patients who achieve R0 resection. For patients with a CY0 status at the time of recruitment, the tumor should be completely removed, and no residual tumor cells within 1 mm of the resection margin should be confirmed by postoperative pathology. For patients with a CY1 status at the time of recruitment, an extra requirement is that CY0 should be confirmed by an peritoneal cytological examination.
Objective response rate (ORR) | 6 months after the recruitment of the last subject.
  The Objective response rate (ORR) is defined as the proportion of patients with a complete response (CR) or a partial response (PR) to preoperative therapy. The ORR will be evaluated using the RESIST1.1 protocol.
Event-free survival (EFS) | 36 months after the recruitment of the last subject.
  The EFS will be calculated from the date of randomization to the date of any event or censoring. The event is defined as below: (1) locoregional recurrence; (2) peritoneal seeding; (3) distant metastasis; (4) death of any reason; (5) tumor progression according to RESIST 1.1.
Overall survival (OS) | 36 months after the recruitment of the last subject.
  The OS will be calculated from the date of randomization to the date of death or date of the last follow-up.
Safety of perioperative therapy include chemo(radio)therapy and PD-1 antibody. | One month after the last date of treatment
  Treatment related adverse events (TRAEs) of perioperative therapy will be graded and documented according to NCI-CTC AE v5.0 from the beginning of treatment to 28 days after the last date of treatment. Documentary will include the occurrence time, severity and time of duration. Common TRAEs include leukopenia, thrombocytopenia, anemia, ALT/AST increase, BUN/Scr increase, nausea, vomiting, diarrhea, appetite decrease, pruritus, rash, fatigue, malaise and pyrexia. Additional TRAEs of special interest include pneumonitis, interstitial lung disease, acute hepatitis, hyperthyroidism, autoimmune thyroiditis, thyroid disorder, hypopituitarism, colitis, maculopapular rash and epidermal capillary hyperplasia.
Safety of surgery after preoperative therapy include chemo(radio)therapy and PD-1 antibody. | During or one month after surgery
  Surgery related adverse events (SRAEs) refer to complications which happen during or one month after surgery. Severe complications after surgery will be documented and classified by Clavien-Dindo grading, such as abdominal or GI tract bleeding, anastomotic fistula, pancreatic fistula of grade B or above, and incision complications (infection, bleeding, rupture).

OTHER OUTCOMES:
To study the association of baseline PD-L1 CPS, TMB, MSI/MMR status, and EBER status on the efficacy of immunotherapy. | 36 months after the recruitment of the last subject.
To study the association between gut microbiota and the efficacy of immunotherapy. | 36 months after the recruitment of the last subject.
To study the association between the Helicobacter pylori infection status and the efficacy of immunotherapy. | 36 months after the recruitment of the last subject.
To study the influence of preoperative therapy on the tumor immune microenvironment (TIME) and systemic immune status. | 36 months after the recruitment of the last subject.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Wang Y, Li Z, Shan F, Miao R, Xue K, Li Z, Gao C, Chen N, Gao X, Li S, Ji J. [Current status of diagnosis and treatment of early gastric cancer in China--Data from China Gastrointestinal Cancer Surgery Union]. Zhonghua Wei Chang Wai Ke Za Zhi. 2018 Feb 25;21(2):168-174. Chinese. PMID 29492915
- [Background] Joshi SS, Badgwell BD. Current treatment and recent progress in gastric cancer. CA Cancer J Clin. 2021 May;71(3):264-279. doi: 10.3322/caac.21657. Epub 2021 Feb 16. PMID 33592120
- [Background] van Hagen P, Hulshof MC, van Lanschot JJ, Steyerberg EW, van Berge Henegouwen MI, Wijnhoven BP, Richel DJ, Nieuwenhuijzen GA, Hospers GA, Bonenkamp JJ, Cuesta MA, Blaisse RJ, Busch OR, ten Kate FJ, Creemers GJ, Punt CJ, Plukker JT, Verheul HM, Spillenaar Bilgen EJ, van Dekken H, van der Sangen MJ, Rozema T, Biermann K, Beukema JC, Piet AH, van Rij CM, Reinders JG, Tilanus HW, van der Gaast A; CROSS Group. Preoperative chemoradiotherapy for esophageal or junctional cancer. N Engl J Med. 2012 May 31;366(22):2074-84. doi: 10.1056/NEJMoa1112088. PMID 22646630
- [Background] Stahl M, Walz MK, Stuschke M, Lehmann N, Meyer HJ, Riera-Knorrenschild J, Langer P, Engenhart-Cabillic R, Bitzer M, Konigsrainer A, Budach W, Wilke H. Phase III comparison of preoperative chemotherapy compared with chemoradiotherapy in patients with locally advanced adenocarcinoma of the esophagogastric junction. J Clin Oncol. 2009 Feb 20;27(6):851-6. doi: 10.1200/JCO.2008.17.0506. Epub 2009 Jan 12. PMID 19139439
- [Background] Leong T, Smithers BM, Haustermans K, Michael M, Gebski V, Miller D, Zalcberg J, Boussioutas A, Findlay M, O'Connell RL, Verghis J, Willis D, Kron T, Crain M, Murray WK, Lordick F, Swallow C, Darling G, Simes J, Wong R. TOPGEAR: A Randomized, Phase III Trial of Perioperative ECF Chemotherapy with or Without Preoperative Chemoradiation for Resectable Gastric Cancer: Interim Results from an International, Intergroup Trial of the AGITG, TROG, EORTC and CCTG. Ann Surg Oncol. 2017 Aug;24(8):2252-2258. doi: 10.1245/s10434-017-5830-6. Epub 2017 Mar 23. PMID 28337660
- [Background] Stahl M, Walz MK, Riera-Knorrenschild J, Stuschke M, Sandermann A, Bitzer M, Wilke H, Budach W. Preoperative chemotherapy versus chemoradiotherapy in locally advanced adenocarcinomas of the oesophagogastric junction (POET): Long-term results of a controlled randomised trial. Eur J Cancer. 2017 Aug;81:183-190. doi: 10.1016/j.ejca.2017.04.027. PMID 28628843
- [Background] Liu X, Jin J, Cai H, Huang H, Zhao G, Zhou Y, Wu J, Du C, Long Z, Fang Y, Ma M, Li G, Zhou M, Yin J, Zhu X, Zhu J, Sheng W, Huang D, Zhu H, Zhang Z, Lu Q, Xie L, Zhang Z, Wang Y. Study protocol of a randomized phase III trial of comparing preoperative chemoradiation with preoperative chemotherapy in patients with locally advanced gastric cancer or esophagogastric junction adenocarcinoma: PREACT. BMC Cancer. 2019 Jun 20;19(1):606. doi: 10.1186/s12885-019-5728-8. PMID 31221115
- [Background] Leong T, Smithers BM, Michael M, Gebski V, Boussioutas A, Miller D, Simes J, Zalcberg J, Haustermans K, Lordick F, Schuhmacher C, Swallow C, Darling G, Wong R. TOPGEAR: a randomised phase III trial of perioperative ECF chemotherapy versus preoperative chemoradiation plus perioperative ECF chemotherapy for resectable gastric cancer (an international, intergroup trial of the AGITG/TROG/EORTC/NCIC CTG). BMC Cancer. 2015 Jul 21;15:532. doi: 10.1186/s12885-015-1529-x. PMID 26194186
- [Background] Slagter AE, Jansen EPM, van Laarhoven HWM, van Sandick JW, van Grieken NCT, Sikorska K, Cats A, Muller-Timmermans P, Hulshof MCCM, Boot H, Los M, Beerepoot LV, Peters FPJ, Hospers GAP, van Etten B, Hartgrink HH, van Berge Henegouwen MI, Nieuwenhuijzen GAP, van Hillegersberg R, van der Peet DL, Grabsch HI, Verheij M. CRITICS-II: a multicentre randomised phase II trial of neo-adjuvant chemotherapy followed by surgery versus neo-adjuvant chemotherapy and subsequent chemoradiotherapy followed by surgery versus neo-adjuvant chemoradiotherapy followed by surgery in resectable gastric cancer. BMC Cancer. 2018 Sep 10;18(1):877. doi: 10.1186/s12885-018-4770-2. PMID 30200910
- [Background] Liu X, Li G, Long Z, Yin J, Zhu X, Sheng W, Huang D, Zhu H, Zhang Z, Cai H, Huang H, Zhao G, Zhou Y, Zhang Z, Wang Y. Phase II trial of preoperative chemoradiation plus perioperative SOX chemotherapy in patients with locally advanced gastric cancer. J Surg Oncol. 2018 Mar;117(4):692-698. doi: 10.1002/jso.24917. Epub 2017 Nov 30. PMID 29194623
- [Background] Zhang X, Liang H, Li Z, Xue Y, Wang Y, Zhou Z, Yu J, Bu Z, Chen L, Du Y, Wang X, Wu A, Li G, Su X, Xiao G, Cui M, Wu D, Chen L, Wu X, Zhou Y, Zhang L, Dang C, He Y, Zhang Z, Sun Y, Li Y, Chen H, Bai Y, Qi C, Yu P, Zhu G, Suo J, Jia B, Li L, Huang C, Li F, Ye Y, Xu H, Wang X, Yuan Y, E JY, Ying X, Yao C, Shen L, Ji J; RESOLVE study group. Perioperative or postoperative adjuvant oxaliplatin with S-1 versus adjuvant oxaliplatin with capecitabine in patients with locally advanced gastric or gastro-oesophageal junction adenocarcinoma undergoing D2 gastrectomy (RESOLVE): an open-label, superiority and non-inferiority, phase 3 randomised controlled trial. Lancet Oncol. 2021 Aug;22(8):1081-1092. doi: 10.1016/S1470-2045(21)00297-7. Epub 2021 Jul 9. PMID 34252374
- [Background] Zhang L, Mai W, Jiang W, Geng Q. Sintilimab: A Promising Anti-Tumor PD-1 Antibody. Front Oncol. 2020 Nov 26;10:594558. doi: 10.3389/fonc.2020.594558. eCollection 2020. PMID 33324564
- [Background] Japanese Gastric Cancer Association. Japanese classification of gastric carcinoma: 3rd English edition. Gastric Cancer. 2011 Jun;14(2):101-12. doi: 10.1007/s10120-011-0041-5. No abstract available. PMID 21573743
- [Background] Japanese Gastric Cancer Association. Japanese gastric cancer treatment guidelines 2014 (ver. 4). Gastric Cancer. 2017 Jan;20(1):1-19. doi: 10.1007/s10120-016-0622-4. Epub 2016 Jun 24. No abstract available. PMID 27342689
- [Background] Oster P, Vaillant L, Riva E, McMillan B, Begka C, Truntzer C, Richard C, Leblond MM, Messaoudene M, Machremi E, Limagne E, Ghiringhelli F, Routy B, Verdeil G, Velin D. Helicobacter pylori infection has a detrimental impact on the efficacy of cancer immunotherapies. Gut. 2022 Mar;71(3):457-466. doi: 10.1136/gutjnl-2020-323392. Epub 2021 Jul 12. PMID 34253574
- [Derived] Zhou M, Yang W, Xuan Y, Zou W, Wang Y, Zhang Z, Zhang J, Mo M, Zhou C, Liu Y, Zhang W, Zhang Z, He Y, Weng W, Tan C, Wang L, Huang D, Sheng W, Li H, Zhu H, Wang Y, Shen L, Zhang H, Wan J, Li G, Huang H, Wang Y, Zhang Z, Liu X, Xia F. A study protocol of a randomized phase II trial of perioperative chemoimmunotherapy verses perioperative chemoimmunotherapy plus preoperative chemoradiation for locally advanced gastric (G) or gastroesophageal junction (GEJ) adenocarcinoma: the NeoRacing study. BMC Cancer. 2022 Jun 28;22(1):710. doi: 10.1186/s12885-022-09786-9. PMID 35764956